CLINICAL TRIAL: NCT07189065
Title: An Open-Label, Randomized Controlled, Multicenter, Phase II Clinical Study to Evaluate the Efficacy and Safety of Rocbrutinib Monotherapy Versus Investigator's Choice of Therapy in Patients With Relapsed or Refractory Non-GCB Diffuse Large B-Cell Lymphoma
Brief Title: A Study of Rocbrutinib in Participants With Relapse or Refractory Non-GCB Diffuse Large B-Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangzhou Lupeng Pharmaceutical Company LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LP-168-CN203
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Diffuse Large B-Cell Lymphoma (DLBCL)
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Bendamustine Hydrochloride; Rituximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rocbrutinib (Experimental)
  Interventions: Drug: Rocbrutinib
- BR/R2 (Active Comparator)
  Interventions: Drug: Bendamustine; Drug: Rituximab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Rocbrutinib — 200mg qd PO. The treatment will continue until progressive disease, unacceptable toxicity, etc.
  Arms: Rocbrutinib
Drug: Bendamustine — Participants will receive a total of 6 cycles (a cycle being 28 days) 90 mg/m2 Bendamustine (IV infusion) on Days 1 and 2 of Cycles 1-6.
  Arms: BR/R2
Drug: Rituximab — Participants will receive a total of 6 cycles (a cycle being 28 days) of 375 mg/m2 Rituximab (IV infusion) on Day 1 of each cycle.
  Arms: BR/R2
Drug: Lenalidomide — 20mg qd PO day 1-21
  Arms: BR/R2

SUMMARY:
This is an open-label, randomized controlled, multicenter Phase II clinical study primarily evaluating the efficacy and safety of Rocbrutinib monotherapy compared to the investigator's choice of BR/R2 regimen in patients with non-GCB DLBCL.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, any gender.
2. Pathologically confirmed DLBCL (not otherwise specified) according to the revised 2017 WHO classification of lymphoid neoplasms, with non-germinal center B-cell-like (non-GCB) subtype confirmed by Han's algorithm (Appendix 1), based on previous pathological records or confirmed during screening. Must be able to provide sufficient tumor tissue or slides (from previous or screening biopsies) for central laboratory confirmation of pathological diagnosis (if the local pathology report is clear, patients may be enrolled and start treatment without waiting for the central pathology report).
3. Patients who are refractory or have relapsed after at least two prior lines of therapy (at least one line must include an anti-CD20 antibody-containing regimen) (see section 6.3 for definition of refractory or relapsed).
4. At least one measurable lesion (nodal lesion with longest diameter >1.5 cm, extranodal lesion with longest diameter >1.0 cm).
5. Not planned for autologous stem cell transplantation (ASCT).
6. Eastern Cooperative Oncology Group (ECOG) performance status score ≤2.

Exclusion Criteria:

1. Primary central nervous system (CNS) lymphoma or known involvement of lymphoma in the CNS (including patients whose CNS lymphoma is currently in complete remission).
2. DLBCL resulting from histological transformation of an previously diagnosed indolent lymphoma [such as follicular lymphoma (FL), marginal zone lymphoma, chronic lymphocytic leukemia, etc.] or pathological findings suggesting concomitant FL (any grade).
3. Diagnosis of other types of large B-cell lymphoma or special types of DLBCL, including but not limited to high-grade B-cell lymphoma, EBV-positive DLBCL, T-cell/histiocyte-rich large B-cell lymphoma, primary mediastinal large B-cell lymphoma, etc.
4. Previous exposure to Lobertinib or known allergy to any excipient of Lobertinib (including microcrystalline cellulose, croscarmellose sodium, magnesium stearate, fumaric acid, and gastric-soluble film coating premix); allergy or intolerance to Rituximab or any of its excipients; allergy or intolerance to both Bendamustine and Lenalidomide or any of their excipients.
5. Previous refractoriness to BTK-targeting drugs.
6. Patients who have received autologous stem cell transplantation within 90 days prior to randomization; patients who have received allogeneic stem cell transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-11-27 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | Up to 24 Months
  To assess the anti-tumor activity of Rocbrutinib and BR/R2 based on overall response rate (ORR) as assessed by Independent Reading Committee (IRC).

SECONDARY OUTCOMES:
Overall Response Rate | Up to 24 Months
  To assess the anti-tumor activity of Rocbrutinib and BR/R2 based on overall response rate (ORR) as assessed by investigator.
Complete remission rate | Up to 24 Months
  To assess the preliminary anti-tumor activity of Rocbrutinib and BR/R2 based on complete remission rate (CR) as assessed by investigator and IRC.
Progression Free Survival | Up to 24 months
  To assess the preliminary anti-tumor activity of Rocbrutinib and BR/R2 based on Progression Free Survival (PFS) as assessed by investigator and IRC.
Overall survival | Measured from the date of date of first dose to the date of death or last visit, and for up to 5 years after the last subject is enrolled.
  To assess the preliminary anti-tumor activity of Rocbrutinib and BR/R2 based on Overall survival (OS) as assessed by investigator and IRC.
Duration of Response (DOR) | Up to 24 months
  To assess the preliminary anti-tumor activity of Rocbrutinib and BR/R2 based on Duration of response (DOR) as assessed by the Investigator and IRC.
Time to Response (TTR) | Measured from the date of the first dose of study drug to the date of earliest response, and assessed up to 6 months.
  To assess the preliminary anti-tumor activity of Rocbrutinib and BR/R2 based on Time to response (TTR) as assessed by the Investigator and IRC.
Safety Assessment | From first dose of study drug to 28 days after last dose of study drug
  To evaluate the safety of Rocbrutinib and BR/R2 by assessing incidence and severity of treatment-emergent adverse events as determined by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (41):
- China (41):
  - Anhui Cancer Hospital (West Branch of Anhui Provincial Hospital), Hefei, Anhui
  - Beijing Shijitan Hospital, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Beijing, Beijing Municipality
  - National Cancer Center/Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Affiliated Cancer Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - Meizhou People's Hospital, Meizhou, Guangdong
  - Affiliated Tumor Hospital of Guangxi Medical University, Nanning, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Affiliated Hospital of Xiamen University, Xiamen, Hujian
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Jilin, Jilin
  - The Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Linyi Cancer Hospital, Linyi, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Shanxi Province Cancer Hospital, Taiyuan, Shanxi
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No